CLINICAL TRIAL: NCT01224548
Title: Multicenter Worksite Nutrition Study
Acronym: WNS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WCCR-WNS2
Record Dates: First submitted 2010-08-30; First posted 2010-10-20 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes; Overweight
Keywords: vegan; diet; diabetes; overweight; workplace; nutrition; diabetes and/or overweight
MeSH Terms: conditions — Diabetes Mellitus; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vegan group (Experimental): participants from sites of this group will receive vegan nutritional intervention starting from Feb 2011
  Interventions: Other: vegan instruction and food accessibility; Other: control
- control group (No Intervention): participants from sites of the control group will not receive the same nutritional information until June 2011

INTERVENTIONS:
Other: vegan instruction and food accessibility — weekly 1-hr instructions including vegan nutritional information and cooking instructions. vegan menu will be made available at the cafeteria
  Arms: vegan group
Other: control — no intervention in until June 2011. The control group start vegan diet in July 2011.
  Arms: vegan group

SUMMARY:
The purpose of this study is to study the potential benefits of low fat vegan diet in a randomized, controlled and multi-centered workplace setting, the investigators will enroll participants from 10 worksites of Government Employee Insurance Company (GEICO). After randomization, 5 will be the vegan sites and 5 will be the control sites for 10 month study. The vegan sites will receive low fat vegan diet instructions and weekly group sessions starting from year 1. no intervention is done to the control sites until the week 18 when the identical program will be given. At various time points, health measurements will be give to all participants.

DETAILED DESCRIPTION:
The purpose of this study is to study the weight loss and other potential benefits of low fat vegan diet as compared to the standard American diet in a randomized, controlled and multi-centered workplace setting.

The 10 months study involves 5 vegan sites and 5 control sites generated through a random process after recruitment. The vegan sites will receive low fat vegan diet instructions and weekly group sessions starting from the January, 2011. The control sites will also receive identical instructions starting from the 5th month and lasting for 18 weeks.

For each participant at baseline and week 18 a blood test will be conducted, along with blood pressure, weight, hip and waist measurements. A questionnaire will also be administered during these time points to assess dietary intake, work productivity, quality of life, and healthcare utilization. At the end of one year, information about health insurance utilization will be obtained from Health Maintenance Organization(HMO) or Preferred Provider Organization(PPO) for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Paid employee at a participating GEICO worksite for at least 6 months
* Currently a full-time employee at GEICO working for GEICO (at least 38.75 hours/week)
* Age of at least 18 years
* Ability and willingness to participate in all components of the study
* A willingness to be assigned to the vegan diet group or the control group
* Body mass index ≥ 25 kg/m2 and/or a diagnosis of type 2 diabetes mellitus, as defined by a fasting plasma glucose concentration ≥ 126 mg/dl on two occasions or a prior physician's diagnosis of type 2 diabetes

Exclusion Criteria:

* A history of alcohol abuse or dependency followed by any current use
* Current or unresolved past drug abuse
* Pregnancy or plans to become pregnant in the next 12 months
* Intention to leave GEICO in the next 12 months
* History of severe mental illness
* Unstable medical status
* Already following a low-fat, vegetarian diet
* An inordinate fear of blood draws
* Previously participated in GEICO two site study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
weight | 0 months
  body weight at baseline
weight | 18 weeks
  body weight at the end of 4 months
weight | 10 months
  body weight at the end of 12 months

SECONDARY OUTCOMES:
blood pressure | 0 months
  diastolic and systolic blood pressures at baseline
blood pressure | 18 weeks
  diastolic and systolic blood pressures at the end of 4 months
blood pressure | 10 months
  diastolic and systolic blood pressures at the end of 12 months
waist circumference | 0 month
  measurement of waist circumference at baseline
waist circumference | 18 weeks
  measurement of waist circumference at 4 months
waist circumference | 10 months
  measurement of waist circumference at 12 months
absenteeism | 0 month
  number of days absent because of sickness over the past 6 months, surveyed at baseline
absenteeism | 18 weeks
  number of days absent because of sickness over the past 4 months, surveyed at the end of 4 months.
absenteeism | 10 months
  number of days absent because of sickness over the past 6 months, surveyed at the end of 12 months.
health insurance utilization | 0 month
  categorized payments by health insurance company for health-related coverage over the past 12 months, surveyed at baseline
healthy insurance utilization | 12 months
  categorized payments by health insurance company for health-related coverage over the past 12 months, surveyed at the end of 12 months
blood lipid panel | 0 month
  blood test of Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), total cholesterol, and triglyceride at baseline
blood lipid panel | 18 weeks
  blood test of Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), total cholesterol, and triglyceride at the end of 4 months
blood lipid panel | 10 months
  blood test of Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), total cholesterol, and triglyceride at the end of 12 months
quality of life | 0 month
  questionnaire on quality of life measurements surveyed at baseline
quality of life | 18 weeks
  questionnaire on quality of life measurements surveyed at the end of 4 months
quality of life | 10 months
  questionnaire on quality of life measurements surveyed at the end of 12 months
hemoglobin A1c | 0 month
  blood test of hemoglobin A1c level (for diabetic participants only) at baseline
hemoglobin A1c | 18 weeks
  blood test of hemoglobin A1c level (for diabetic participants only) at the end of 4 months
hemoglobin A1c | 10 months
  blood test of hemoglobin A1c level (for diabetic participants only) at the end of 12 months
hip circumference | 0 month
  measurement of hip circumference at baseline
hip circumference | 18 weeks
  measurement of hip circumference at the end of 4 months
hip circumference | 10 months
  measurement of hip circumference at the end of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, M.D., Principal Investigator — Washington Center for Clinical Research
Locations (10):
- United States (10):
  - Tucson, Tucson, Arizona
  - San Diego, San Diego, California
  - Lakeland, Lakeland, Florida
  - Macon, Macon, Georgia
  - Chevy Chase, Chevy Chase, Maryland
  - Buffalo, Buffalo, New York
  - Woodbury, Woodbury, New York
  - Dallas, Dallas, Texas
  - Fredericksburg, Fredericksburg, Virginia
  - Virginia Beach, Virginia Beach, Virginia